CLINICAL TRIAL: NCT00467805
Title: Immediate Effect of Light on Reproductive Hormones in Women: a Role of the Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Outside In
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: M-s4c
Record Dates: First submitted 2007-04-30; First posted 2007-05-01 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2009-10

CONDITIONS: Healthy
Keywords: Light exposure; light spectrum; reproductive hormones; women
MeSH Terms: interventions — Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Light therapy

SUMMARY:
The study investigates an acute effect of white-appearing LED light (with a peak in blue portion) vs. red LED light of similar irradiance on reproductive hormones in healthy women.

DETAILED DESCRIPTION:
Sixteen healthy women came to the laboratory at 7:30 (wearing dark goggles) at two occasions (separated by 2-3 days, first time - at the 3rd-8th day of their menstrual cycle) to be exposed for 45' to white-appearing or red LED light (sequential allocation). The white light has a distinct peak at 460 nm, the narrow-band red light peaked at 651 nm. The LED devices were positioned at the distance of 50 cm (white) and 45 cm (red) from the eyes to be matched by irradiance (approximately 7.0 microWt/m2); background light in direction of gaze was 5-10 lux. Blood and saliva samples were collected before, in the middle, and during the last minutes of the 45' exposure to be measured later for concentration of luteinizing hormone, follicle-stimulating hormone, prolactin, estrogen, progesterone, and also - for cortisol and melatonin (the last one - in saliva) as well-studied indicators of the direct effect of light.

ELIGIBILITY:
Inclusion Criteria:

* age 18-45 y
* normal (21-35 days) menstrual cycle
* good and stable general health
* normal body weight index 18.5-29.9
* normal sleep-wake regimen
* living close to the laboratory (<7' by walk)
* "good"cubital veins

Exclusion Criteria:

* difficulty to contact
* travel over several time zones during last month
* medications known to interfere with hormone release

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Reproductive hormones concentration | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin V Danilenko, MD, Study Chair — Institute of Internal Medicine SB RAMS; Oksana Y. Sergeeva, PhD student, Principal Investigator — Institute of Internal Medicine SB RAMS
Locations (1):
- Institute of Internal Medicine SB RAMS, Novosibirsk, Russia